CLINICAL TRIAL: NCT04707053
Title: Data Collection and Analysis of Neuroimaging and Intraoperative Neurophysiological Monitoring (IONM) in Brainstem Surgeries
Brief Title: Data Collection and Analysis in Brainstem Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yang Yang, MD, Dr., Cantonal Hospital of St. Gallen
Other Study IDs: 2020-02088
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Brainstem Lesion; Surgery; Intraoperative Neurophysiologic Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intraaxial lesion group: Patients with intraaxial brainstem lesions (lesions located in the brainstem) + experienced brainstem surgery in our department during the study period
- Extraaxial lesion group: Patients with extraaxial brainstem lesions (lesions close to the brainstem) + experienced brainstem surgery in our department during the study period

SUMMARY:
The hypothesis is that the structural documentation and analysis of the data of demographics, neuroimaging, IONM and clinical outcomes can help to further standardize the use of such equipment for detecting the integrity of the corticospinal tracts.

We want to confirm that the retrospectively data analysis of neuroimaging, IONM and clinical outcomes does help to understand these methods better in the surgical management of brainstem lesions, and therefore, improve the safety of brainstem surgery.

DETAILED DESCRIPTION:
This will be a prospective data collection and retrospective data analysis study to investigate the effect of pre- and post-neuroimaging, intraoperative monitoring, and clinical outcome during the surgical management of brainstem lesions in our neurosurgical center. The data of demographics, neuroimaging, IONM and patients' outcomes will be acquired based on the medical records and follow-up visits. All data is stored in the personal file of the clinical information system for each patient. The expected duration of each subject's participation is confined to the surgery itself and the routine visits during the follow-up. The overall study duration is expected to collect all the brainstem surgery in next five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 80 years' old
* With lesions in or near the brainstem
* Patients who are suitable for brainstem surgery
* Patients who accept the surgery
* Patients who signed the informed consent

Exclusion Criteria:

* Patients age < 18 years
* Patients who are not suitable for brainstem surgery (for example patients in coma, very small lesion, pregnancy)
* Patients unlikely to attend the follow-up 12 months after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with lesions in or near brainstem who accept surgical resection as the optimal treatment. Estimation of 50 participants in the intra-axial brainstem surgical group, and 150 in the extra-axial brainstem surgical group. There is no other patient collective that could be used as substitute for the study population.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Data of direct brainstem stimulation and clinical outcome | 09/2020-12/2021
  The measurement of stimulation intensity (in mA) and its corresponding neurophysiological outcome (positive or not), as well as the short- and long-term neurological outcome (mRS 0-6) help the standardization of direct brainstem stimulation and clinical outcome prediction

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bozinov, Prof, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland